CLINICAL TRIAL: NCT05899998
Title: Bright IDEAS for Pediatric Palliative Care: A Problem-Solving Skills Intervention to Empower Parent Resilience
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Los Angeles (Other)
Responsible Party: Principal Investigator, Bemis, Heather, Principal Investigator, Children's Hospital Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CHLA-23-00162
Record Dates: First submitted 2023-05-26; First posted 2023-06-12 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Psychological Distress; Quality of Life
Keywords: Depressive Symptoms; Anxiety; Post-Traumatic Stress
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bright IDEAS (Experimental)
  Interventions: Behavioral: Bright IDEAS
- Standard of Care (No Intervention)

INTERVENTIONS:
Behavioral: Bright IDEAS — Bright IDEAS® (Identify, Define, Evaluate, Act, See) is a problem-solving skills training program that was originally developed to alleviate distress in caregivers of children recently diagnosed with cancer. Intervention materials include instructor and user manuals, a brochure, and worksheets to be completed by the parent caregiver, initially with the help of the interventionist and then with increasing independence.
  Arms: Bright IDEAS

SUMMARY:
The goal of this or clinical trial is to test in the feasibility, acceptability and preliminary efficacy of the bright IDEAS problem solving skills training for parents of children in palliative care. The main questions it aims to answer are:

* Is bright IDEAS problem solving skills training feasible and acceptable for parents of children referred to pediatric palliative care?
* Does bright IDEAS reduce psychological distress in parents compared to parents receiving standard palliative care support?

Participants will:

* Participate in 6-8 sessions of the bright IDEAS program.
* Complete self report measures of psychological distress and well being.

If there is a comparison group: Researchers will compare bright IDEAS to standard palliative care support.

ELIGIBILITY:
Parent

Inclusion Criteria:

* Parents or legal guardians of male and female children (ages 0-21) of any race or ethnicity and of any underlying medical diagnosis
* Child received at least one consult from the Comfort and Palliative Care team within the past month
* One parent or primary caregiver per child
* Able to speak, read, and write English or Spanish, and give informed consent

Exclusion Criteria:

* Parent age less than 18 years old
* Concurrent enrollment on another research study testing psychoeducational interventions for parents and/or patients
* Child has an estimated life expectancy of less than 4 months at time of study recruitment

Child

Inclusion Criteria:

* Children 8-17 years of age whose primary caregiver has consented to participate
* Able to read and write English or Spanish and assent

Exclusion Criteria:

• Parent refusal to participate

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-08-08 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Feasibility of Bright IDEAS for parents | Baseline to 12 weeks
  Percent eligible participants who consent/assent to participate and Number of sessions completed by enrolled participants.
Parent Problem-Solving skills | Baseline to 16 weeks
  Social Problem-Solving Inventory-Revised Short Form. This is a a 25-item self-report instrument that measures five dimensions of problem-solving (positive problem orientation, negative problem orientation, rational problem-solving style, impulsive/carelessness style, and avoidant style) using a five-point Likert scale (0 = "Not at All True of Me" to 4 = "Extremely True of Me"). Summary scores for each subscale as well as a Total Raw Score range from 0-20. Higher scores indicate better self-reported problem-solving skills.
Anxiety symptoms | Baseline to 16 weeks
  PROMIS® Anxiety Short Form-v1.0 8a. This self-report measure includes includes 8 items on which participants respond using a 5-point scale (1 = "Never" to 5 = "Always"). Total raw scores range from 8-40 and are converted to standardized T-scores with a mean of 50 and standard deviation of 10. Higher scores indicate higher levels of anxiety.
Depression symptoms | Baseline to 16 weeks
  PROMIS® Depression Short Form-v 1.0 8a. This self-report measure includes includes 8 items on which participants respond using a 5-point scale (1 = "Never" to 5 = "Always"). Total raw scores range from 8-40 and are converted to standardized T-scores with a mean of 50 and standard deviation of 10. Higher scores indicate higher levels of depressive symptoms.
Traumatic stress symptoms | Baseline to 16 weeks
  Abbreviated Posttraumatic Checklist -Civilian Version (PCL-6). This is a 6-item self-report screening measure empirically derived from the PCL-C, consisting of the most highly responsive items from each of the reexperiencing, avoidance, and hyperarousal symptom domains of the PCL-C and has previously been used with parents of children with serious illness. The PCL-6 uses a five-point Likert scale (0 = "Not at all" to 5 = "Extremely"), with total scores ranging from 6-30. Higher scores indicate higher levels of traumatic stress symptoms.

SECONDARY OUTCOMES:
Parent Wellbeing | Baseline to 16 weeks
  CarerQoL. The CarerQOL evaluates care-related quality of life and incorporates caregiving burden as well as positive effects of caregiving. It consists of 7 items related to caregiving burdens, fulfillment, or support that participants self-rate on a 3-point qualitative scale ("No", "Some" or "A lot of") as well as 1 item in which the respondent rates their current overall happiness on a 10-point visual analog scale with higher scores corresponding to higher positive affect (0 = "completely unhappy" to 10 = "completely happy"). The measure will be slightly adapted to clarify reference to the child as the care receiver.
Child Quality of Life (QoL) Parent Proxy 0-7 years old | Baseline to 16 weeks
  PROMIS® Early Childhood Parent Report Global Health 8a contains 8 items, assessing global health and development. All items use a 5-point Likert scale (1 = Poor to 5 = Excellent). Total raw sum scores range from 8-40 and are converted to standardized T-scores with a mean of 50 and standard deviation of 10. Higher scores indicate better reported wellbeing.
Child Quality of Life (QoL) Parent Proxy 8+ years old | Baseline to 16 weeks
  PROMIS® Parent Proxy Scale v1.0 Global Health 7+2. This measure contains 9 items in total, including 7 items assessing global health (physical and mental wellbeing), and 1 item each related to fatigue and pain burden. All items are completed on a 5-point Likert scale (anchors are 1= Poor to 5 = Excellent, or 1 = Never to 5 = Always or Almost always, depending on the domain). Total raw sum scores for global health range from 7-35 and are converted to standardized T-scores with a mean of 50 and standard deviation of 10. Raw scores for the fatigue and pain items each range from 1-4 and are each separately converted to standardized T-scores with a mean of 50 and standard deviation of 10. Higher scores indicate better reported wellbeing and lower fatigue and pain, respectively.
Child Quality of Life (QoL) Child Self-Report | Baseline to 16 weeks
  Participating parents' child (ages 8+) who are medically and cognitively able will be invited to complete the PROMIS® Pediatric Scale v1.0 Global Health 7+2 to measure self-reported quality of life. This measure contains 9 items in total, including 7 items assessing global health (physical and mental wellbeing), and 1 item each related to fatigue and pain burden. All items are completed on a 5-point Likert scale (anchors are 1= Poor to 5 = Excellent, or 1 = Never to 5 = Always or Almost always, depending on the domain). Total raw sum scores for global health range from 7-35 and are converted to standardized T-scores with a mean of 50 and standard deviation of 10. Raw scores for the fatigue and pain items each range from 1-4 and are each separately converted to standardized T-scores with a mean of 50 and standard deviation of 10. Higher scores indicate better reported wellbeing and lower fatigue and pain, respectively.

OTHER OUTCOMES:
Bright IDEAS Acceptability | Between Time 2 and Time 3, up to 16 weeks
  Qualitative Interviews will assess participant satisfaction with the intervention format, timing, and content; impact; barriers; and suggestions for refinement.

CONTACTS AND LOCATIONS:
Overall Officials: Heather Bemis, PhD, Principal Investigator — Children's Hospital Los Angeles
Locations (1):
- Children's Hospital Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No